CLINICAL TRIAL: NCT02733263
Title: Resistant Maltodextrin Supplementation and the Effect on Fecal Bifidobacteria, Bowel Function, Dietary Intake and Quality of Life
Brief Title: Resistant Maltodextrin Supplementation: Gastrointestinal Health
Acronym: DEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: ADM/Matsutani LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB201501168
Record Dates: First submitted 2016-03-25; First posted 2016-04-11 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: gut microbiota; fiber; diet quality; immunity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Participants will first consume in the the order of 0 g RMD, 15 g RMD, 25 g RMD for 3 weeks each
  Interventions: Dietary Supplement: 15 g RMD; Dietary Supplement: 25 g RMD; Dietary Supplement: 0 g RMD
- Group 2 (Experimental): Participants will first consume RMD in the the order of 0 g RMD, 25 g RMD, 15 g RMD for 3 weeks each
  Interventions: Dietary Supplement: 15 g RMD; Dietary Supplement: 25 g RMD; Dietary Supplement: 0 g RMD
- Group 3 (Experimental): Participants will first consume RMD in the the order of 15 g RMD, 0 g RMD, 25 g RMD for 3 weeks each
  Interventions: Dietary Supplement: 15 g RMD; Dietary Supplement: 25 g RMD; Dietary Supplement: 0 g RMD
- Group 4 (Experimental): Participants will first consume RMD in the the order of 15 g RMD, 25 g RMD, 0 g RMD for 3 weeks each
  Interventions: Dietary Supplement: 15 g RMD; Dietary Supplement: 25 g RMD; Dietary Supplement: 0 g RMD
- Group 5 (Experimental): Participants will first consume RMD in the the order of 25 g RMD, 15 g RMD, 0 g RMD for 3 weeks each
  Interventions: Dietary Supplement: 15 g RMD; Dietary Supplement: 25 g RMD; Dietary Supplement: 0 g RMD
- Group 6 (Experimental): Participants will first consume RMD in the the order of 25 g RMD, 0 g RMD, 15 g RMD for 3 weeks each
  Interventions: Dietary Supplement: 15 g RMD; Dietary Supplement: 25 g RMD; Dietary Supplement: 0 g RMD

INTERVENTIONS:
Dietary Supplement: 15 g RMD — 15 grams of resistant maltodextrin
Dietary Supplement: 25 g RMD — 25 grams of resistant maltodextrin
Dietary Supplement: 0 g RMD — 0 grams of resistant maltodextrin

SUMMARY:
Resistant maltodextrin (RMD) is an indigestible water soluble fiber that increases fecal bulk by enhancing growth of specific microbial populations; however the effect of RMD on bifidobacteria and total fecal weight is not clear. The purpose of this research study is to determine whether incorporating about ¼ cup of a fiber supplement into the diet will induce beneficial changes in gastrointestinal function, the fecal microbiota profile (increased number of healthy bacteria in stool) and immune processes resulting in improved quality of life.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. After obtaining informed consent, participants will be randomized to either consume 0, 15 or 25 grams of resistant maltodextrin (RMD) during the first arm of the study. During the first intervention period, participants will consume the RMD everyday for 3 weeks. After a 2-week post intervention period, participants will be crossed to one of the other treatments for 3 weeks, followed by a 2-week post intervention and then receive the final intervention for 3 weeks.

Participants will complete daily questionnaires and weekly gastrointestinal symptom questionnaires during the intervention and post-intervention periods. Stool samples will be collected at the baseline and final time points of each intervention. Dietary intake will also be assessed weekly during each intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.5 to <30 kg/m2
* Usual fiber intake of <19 g/d for males and 13 g/d for females based on Food Frequency Questionnaire (FFQ) such as the NutritionQuest Fruit/Vegetable/Fiber Screener.
* Willing to complete daily and weekly questionnaires, 20 dietary recalls, and 15 stool collection days over approximately 18 weeks
* Willing to drink the study supplements for 3 weeks for each of the three intervention periods
* Willing to discontinue any prebiotic, fiber, or probiotic supplements or foods containing probiotics (e.g., yogurts with live, active cultures)
* Internet access for the duration of the protocol to complete online questionnaires
* On average you have 6 or more stools but fewer than 12

Exclusion Criteria:

* Does not meet above criteria
* Dietary fiber intake greater than half the adequate intake (AI) based on Automated Self-Administered Diet History (ASA24) (http://riskfactor.cancer.gov/tools/instruments/asa24/) dietary intake data collected during run-in period:

  * Females with a dietary fiber ≥13 g/d
  * Males with a dietary fiber ≥19 g/d
* Antibiotic use within 2 months from providing the screening stool sample
* Physician-diagnosed gastrointestinal disease or condition (such as ulcerative colitis, Crohn's disease, gastroparesis, cancer, peptic ulcer disease, Celiac disease, short bowel disease, ileostomy, colostomy) other than Gastroesophageal Reflux Disease (GERD), constipation, or diverticular disease
* Purposeful strenuous exercise of >300 minutes per week on average
* Women who are lactating or know they are pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06-30 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Fecal bifidobacteria counts | Baseline (Week 0) and Final (Week 3) of each intervention
  The mean of the change between baseline and final time points in stool bifidobacteria counts [log(CFU)] was compared for each study arm.

SECONDARY OUTCOMES:
Fecal weight | Baseline (Week 0) and Final (Week 3) of each intervention
  Average stool weight and consistency for each intervention
Gastrointestinal Function as a measure of changes in average number of stools | Baseline (Week 0) and Final (Week 3) of each intervention
  Changes in average number of stools per week were measured using a Daily Questionnaire. Results were compared between treatment periods for each subject/group.
Immune Status by biomarker sIgA | Baseline (Week 0) and Final (Week 3) of each intervention
  Marker or immune status Secretory Immunoglobulin A (sIgA) using sIgA ELISA
Diet Quality | Week 3 of each intervention
  Six dietary recalls occurred per study intervention, and each recall was scored for quality. The quality scores were averaged per arm and then compared between study arms for each subject/group using the Healthy Eating Index-2010.The Healthy Eating Index assesses diet quality based on 12 components, when summed has maximum points of 100 (HEI scale 0-100).
  High component scores indicate intakes close to the recommended ranges or amounts; low component scores indicate less compliance with the recommended ranges or amounts.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No